CLINICAL TRIAL: NCT02719600
Title: Motor Learning Through Virtual Reality Task in Individuals With Down Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Carlos Bandeira de Mello Monteiro, Professor, University of Sao Paulo
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1033/03
Record Dates: First submitted 2016-03-03; First posted 2016-03-25 (Estimated); Last update posted 2016-03-25 (Estimated); Status verified 2016-03

CONDITIONS: Down Syndrome
Keywords: Virtual Reality
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Down Syndrome Group (Experimental): Group with Down Syndrome
  Interventions: Behavioral: Virtual reality
- Typical Development Group (Active Comparator): Control group with typical development
  Interventions: Behavioral: Virtual reality

INTERVENTIONS:
Behavioral: Virtual reality — Evaluation of observational motor learning using virtual reality

SUMMARY:
Background: Down syndrome (DS) has unique physical, motor and cognitive characteristics. Despite cognitive and motor difficulties, there is a possibility of intervention based on the knowledge of motor learning. However, it is important to study the motor learning process in individuals with DS during a virtual reality task to justify the use of virtual reality to organize intervention programs. The aim of this study was to analyze the motor learning process in individuals with DS during a virtual reality task. Methods: A total of 40 individuals participated in this study, 20 of which were with DS (24 males and 8 females, ranging between 11-28 yrs.) and 20 typically developing individuals matched by age and gender to the individuals with DS. To examine this issue, we used software that uses 3D images and reproduced a coincidence timing task.

ELIGIBILITY:
Inclusion Criteria:

* medical diagnosis of DS and the ability to understand the task.

Exclusion Criteria:

* disorders in cognitive function that would prevent comprehension of the experimental instruction

Ages: 11 Years to 28 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2015-03; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Motor Learning test by using a timing coincident task in virtual reality | four months
  Improvement on their performance, by reaching the task with precision

CONTACTS AND LOCATIONS:
Overall Officials: Carlos B Monteiro, PhD., Principal Investigator — University of Sao Paulo

IPD SHARING:
Plan to Share IPD: No
No interest on sharing individual participant data

REFERENCES:
- [Derived] de Mello Monteiro CB, da Silva TD, de Abreu LC, Fregni F, de Araujo LV, Ferreira FHIB, Leone C. Short-term motor learning through non-immersive virtual reality task in individuals with down syndrome. BMC Neurol. 2017 Apr 14;17(1):71. doi: 10.1186/s12883-017-0852-z. PMID 28410583